CLINICAL TRIAL: NCT01236196
Title: Telephone Cognitive Behavior Therapy for OEF Veterans With Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D7658-I
Record Dates: First submitted 2010-11-01; First posted 2010-11-08 (Estimated); Results first posted 2014-12-23 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Pain
Keywords: pain; chronic pain; cognitive therapy; telehealth
MeSH Terms: conditions — Chronic Pain; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 - Telephone CBT (Experimental): telephone cognitive behavior therapy for pain management
  Interventions: Behavioral: Telephone cognitive behavior therapy
- Arm 2 - telephone education (Active Comparator): telephone pain education
  Interventions: Behavioral: Telephone pain education

INTERVENTIONS:
Behavioral: Telephone cognitive behavior therapy — Cognitive behavior therapy aimed at teaching pain coping skills was conducted by telephone (12 sessions over a 6-month period).
  Arms: Arm 1 - Telephone CBT
Behavioral: Telephone pain education — Participants received information on the management of chronic pain during 12 telephone sessions conducted over a 6-month period).
  Arms: Arm 2 - telephone education

SUMMARY:
We conducted a randomized clinical trial comparing telephone-delivered cognitive behavior therapy and pain education control. We enrolled 41 OEF/OIF/OND veterans with chronic pain and randomizing them into one of two treatment conditions. The study sample was recruited from primary care clinics at the San Francisco VA Medical Center and affiliated VA community-based outpatient clinics (CBOCs) in downtown San Francisco, Clearlake, Eureka, San Bruno, Santa Rosa, and Ukiah. Recruitment targeted OEF/OIF/OND veterans with pain disorders that involved muscle strain and inflammation, trauma to nerves, and/or central nervous system dysfunction. Both interventions were delivered by telephone and consisted of 12 sessions scheduled over a 20-week period. Pain management outcomes were measured at 10 weeks (mid-treatment), 20 weeks (post-treatment), 32 weeks (3-month follow-up), and 46 weeks (6-month follow-up). The sample size was chosen to provide greater than 80% power at a two-tailed alpha of 0.05. The study hypothesis, assessment methodology, and intervention procedures were based on the cognitive-behavioral model of chronic pain.

DETAILED DESCRIPTION:
In the VHA, over 50% of OEF/OIF/OND veterans who are seen in primary care settings report disabling pain symptoms. Although cognitive behavior therapy (CBT) is now commonly employed within interdisciplinary pain management programs, access to these interventions is often limited due to the distance from clinical care and disabling impact of pain. In addition, the dropout rate in studies of face-to-face CBT for chronic pain further detracts from its impact in pain management. A telephone-delivered version of CBT for chronic pain overcomes these barriers to access.

Primary Aim: to investigate the effectiveness of telephone CBT in the management of chronic pain with OEF/OIF/OND veterans enrolled in VA primary care clinics.

Secondary Aim: to determine moderator and mediating factors by which telephone CBT facilitates pain management and successful adjustment of OEF/OIF/OND veterans to chronic pain.

Major hypothesis:

Hypothesis 1: Patients who receive telephone CBT will show significantly greater improvements in coping skills, reduced emotional distress, and increased quality of life compared with those who participate in telephone pain education (EDU).

Hypothesis 2: The dropout rate for both of the telephone interventions in this study will be significantly lower than the attrition rate found in previous studies of face-to-face CBT for chronic pain.

Secondary hypothesis:

Hypothesis 3: An increase in use of coping skills will be positively associated with treatment outcome measures reflecting improved adjustment to chronic pain.

Hypothesis 4: A decrease in catastrophizing will be positively associated with treatment outcome measures reflecting improved adjustment to chronic pain.

To accomplish these aims, we conducted a randomized clinical trial comparing telephone-delivered cognitive behavior therapy and pain education control. A total of 42 OEF/OIF/OND veterans with chronic pain were enrolled in the study and randomized into one of two treatment conditions. The study sample was recruited from primary care clinics at the San Francisco VA Medical Center and affiliated VA community-based outpatient clinics (CBOCs) in downtown San Francisco, Eureka, San Bruno, Santa Rosa, and Ukiah. Recruitment targeted OEF/OIF/OND veterans with pain disorders that involved muscle strain and inflammation, trauma to nerves, and/or central nervous system dysfunction. Both interventions were delivered by telephone and consisted of 12 sessions scheduled over a 20-week period. Pain management outcomes were measured at 10 weeks (mid-treatment), 20 weeks (post-treatment), 32 weeks (3-month follow-up), and 46 weeks (6-month follow-up). The sample size was chosen to provide greater than 80% power at a two-tailed alpha of 0.05. The study hypothesis, assessment methodology, and intervention procedures were based on the cognitive-behavioral model of chronic pain.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, potential subjects must have:

* access to a telephone
* documented pain for at least the past year
* a pain disorder involving muscle strain and inflammation, trauma to nerves, or central nervous system dysfunction
* pain condition must be stable
* must have no clear indication for specific medical/surgical intervention.

Exclusion Criteria:

Patients were excluded who were:

* acutely psychotic
* cognitively impaired
* showed significant suicidal risk (history of multiple suicide attempts or actively suicidal)
* currently abusing alcohol or other drugs, including prescribed opioid pain medications
* patients were also excluded who had an unstable medical condition and clear indication for specific medical/surgical intervention in the near future.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2010-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Carmody, PhD, Principal Investigator — VA Medical Center, San Francisco
Locations (1):
- VA Medical Center, San Francisco, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 41 veterans were enrolled, but 2 dropped out before being randomized to treatment condition and did not receive either treatment.
Period: Overall Study
Arm/Group | Arm 1 - Telephone CBT | Arm 2 - Telephone Education
Started | 18 | 21
Completed | 17 | 13
Not Completed | 1 | 8

BASELINE CHARACTERISTICS:
Population: OEF/OIF/OND military veterans with chronic pain
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 - Telephone CBT | Arm 2 - Telephone Education | Total
Number analyzed (Participants) | 18 | 21 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (11) | 34 (10) | 35 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 16 | 16 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 16 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 5 | 16
Region of Enrollment [Number; unit: participants]
  United States | 18 | 21 | 39
Marital status [Number; unit: participants]
  Married | 5 | 7 | 12
  Not married | 13 | 14 | 27
Education [Mean (Standard Deviation); unit: years] | 15 (2) | 15 (2) | 15 (2)

OUTCOME MEASURES:

1. Primary Outcome: Level of Functioning
Description: Physical health (quality of life), reported on the SF-12, range 0-100, higher scores reflect better quality of life and higher level of functioning
Time Frame: Baseline, 46 weeks
Population: OEF/OIF/OND military veterans with chronic pain
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 - Telephone CBT | Arm 2 - Telephone Education
Number analyzed (Participants) | 18 | 21
units on a scale
  46 weeks | 47 (11) | 37 (12)
  Baseline | 41 (12) | 36 (9)
Statistical Analysis 1: Comparison: Arm 1 - Telephone CBT vs Arm 2 - Telephone Education; Test type: Superiority or Other; p = 0.11, Mixed Models Analysis

2. Primary Outcome: Depressive Symptoms
Description: Depressive symptoms, measured on Beck Depression Inventory-II (total score with range from 0 to 63)
Time Frame: Baseline, 46 weeks
Population: OEF/OIF/OND military veterans with chronic pain
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 - Telephone CBT | Arm 2 - Telephone Education
Number analyzed (Participants) | 18 | 21
units on a scale
  46 weeks | 12 (11) | 12 (10)
  Baseline | 13 (8) | 18 (13)
Statistical Analysis 1: Comparison: Arm 1 - Telephone CBT vs Arm 2 - Telephone Education; Test type: Superiority or Other; p = 0.80, Mixed Models Analysis

3. Primary Outcome: Pain Behavior
Description: Pain behavior measured as total score on Pain Behavior Checklist (range 0-6), higher score indicating more pain behavior
Time Frame: Baseline, 46 weeks
Population: OEF/OIF/OND military veterans with chronic pain
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 - Telephone CBT | Arm 2 - Telephone Education
Number analyzed (Participants) | 18 | 21
units on a scale
  46 weeks | 1.0 (1.0) | 2.1 (1.4)
  Baseline | 1.2 (1) | 2.4 (1)
Statistical Analysis 1: Comparison: Arm 1 - Telephone CBT vs Arm 2 - Telephone Education; Test type: Superiority or Other; p = 0.01, Mixed Models Analysis

4. Primary Outcome: Pain Intensity
Description: Pain Intensity Rating, ranging from 0-6, higher score indicates greater pain intensity
Time Frame: Baseline, 46 weeks
Population: OEF/OIF/OND military veterans with chronic pain
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 - Telephone CBT | Arm 2 - Telephone Education
Number analyzed (Participants) | 18 | 21
units on a scale
  46 weeks | 3.1 (2.2) | 4.8 (2.6)
  Baseline | 3.2 (1.9) | 5.6 (2.3)
Statistical Analysis 1: Comparison: Arm 1 - Telephone CBT vs Arm 2 - Telephone Education; Test type: Superiority or Other; p = 0.09, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 46 weeks
Arm/Group | Arm 1 - Telephone CBT | Arm 2 - Telephone Education
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/21
Other Adverse Events (participants affected / at risk) | 0/18 | 0/21

LIMITATIONS AND CAVEATS:
The fact that this study was conducted in northern California may have posed some threat to external validity when applying these findings to the nationwise VA system.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No